CLINICAL TRIAL: NCT05687318
Title: A Clinical Trial of the Effectiveness and Safety of Software Assisting Diagnose the Intestinal Polyp Digestive Endoscopy by Analysis of Colonoscopy Medical Images From Electronic Digestive Endoscopy Equipment, a Prospective, Multicenter, Randomized Stratified Block, Incomplete Blind Setting, Parallel Sequential Control, and Efficacy Test
Brief Title: A Clinical Trial of the Effectiveness and Safety of Software Assisting Diagnose the Intestinal Polyp Digestive Endoscopy by Analysis of Colonoscopy Medical Images From Electronic Digestive Endoscopy Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Second Hospital University of South China (Other); Loudi Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: PekingUMCH-1
Record Dates: First submitted 2023-01-03; First posted 2023-01-18 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2022-12

CONDITIONS: Artificial Intelligence; Enteroscope; Intestinal Polyposis, Adenomatous
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Ⅰ (Experimental): Subjects underwent colonoscopy with the investigator's combined instrument, and then underwent traditional colonoscopy with the same investigator
  Interventions: Device: DeFrame
- Trial Ⅱ (Experimental): Subjects underwent a traditional colonoscopy, followed by a colonoscopy with the same investigator's instrument
  Interventions: Device: DeFrame

INTERVENTIONS:
Device: DeFrame — DeFrame can analyze colonoscopy medical images generated by electronic digestive endoscopy equipment to automatically identify, label and screen capture polyps in the colon.

SUMMARY:
A clinical trial of the effectiveness and safety of intestinal polyp digestive endoscopy-assisted diagnosis software used in the analysis of colonoscopy medical images generated by electronic digestive endoscopy equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 85 years old, regardless of gender;
* electronic colonoscopy is required;
* The subjects or their legal representatives could understand the purpose of the trial, show sufficient compliance with the trial protocol, and sign the informed consent.

Exclusion Criteria:

* (1) Contraindications associated with electronic colonoscopy or biopsy;
* (2) poor intestinal preparation;
* (3) diagnosed colorectal cancer, familial polyposis, or complicated with known colorectal polyps;
* (4) serious neurological diseases or dysfunction of vital organs (heart, lung, liver, kidney);
* (5) acute abdominal or intestinal inflammation;
* (6) History of abdominal, pelvic, anal and perianal operations within 2 months before enrollment;
* (7) Participated in other interventional clinical trials within 1 month before enrollment;
* (8) In the interest of subjects, the investigator considers that they should not participate in other conditions of the clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
PMR | during colonoscopy procedure
  Polyp miss rate

SECONDARY OUTCOMES:
AMR | during colonoscopy procedure
  Adenoma miss rate

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No